CLINICAL TRIAL: NCT04825964
Title: Comparison of Exercise Capacity and Physical Activity Levels in Patients With Hyperthyroid and Healthy Controls
Brief Title: Exercise Capacity, Physical Activity Levels in Patients With Hyperthyroid
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi University 25
Record Dates: First submitted 2021-03-20; First posted 2021-04-01 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Hyperthyroidism
Keywords: Hyperthyroidism; Exercise Capacity; Physical Activity
MeSH Terms: conditions — Hyperthyroidism; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Functional exercise capacity (6 minutes walk test and 6 minutes stepper test), physical activity level (multi-sensor activity monitor), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), peripheral muscle strength (dynamometer), respiratory muscle endurance (incremental threshold loading test), quality of life (The Thyroid-Related Quality of Life-ThyPRO), fatigue (Fatigue Severity Scale), depression-anxiety-stress (Depression Anxiety Stress Scale-42), quality of sleep (Pittsburgh Sleep Quality Index) and shortness of breath (Modified Medical Research Council (MMRC)) will be evaluated at diagnosis and after 1-3 months.
- Healthy Controls: Functional exercise capacity (6 minutes walk test and 6 minutes stepper test), physical activity level (multi-sensor activity monitor), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), peripheral muscle strength (dynamometer), respiratory muscle endurance (incremental threshold loading test), quality of life (The Thyroid-Related Quality of Life-ThyPRO), fatigue (Fatigue Severity Scale), depression-anxiety-stress (Depression Anxiety Stress Scale-42), quality of sleep (Pittsburgh Sleep Quality Index) and shortness of breath (Modified Medical Research Council (MMRC)) will be evaluated one time.

SUMMARY:
The primary aim of the study is to evaluate physical activity level and functional exercise capacity in patients with hyperthyroid. The secondary aim of the study is assessment of respiratory function, peripheral and respiratory muscle strength, respiratory muscle endurance, fatigue, depression, anxiety, stress, sleep and quality of life in patients with hyperthyroid and compare them with healthy controls.

DETAILED DESCRIPTION:
Hyperthyroidism is a pathological disease in which the synthesis and secretion of thyroid hormones are increased by the thyroid gland. Thyroid hormone excess affects many systems. Common clinical symptoms are fatigue, palpitations, disturbed sleep, weight loss, heat intolerance, sweating, tremors, polydipsia, and anxiety. Common physical findings are tachycardia, extremity tremors and weight loss.

Thyroid hormone directly affects skeletal muscles. Increased thyroid hormone causes myopathy with a decrease in muscle strength and mass. Hyperthyroid myopathy can cause a decrease in exercise capacity. The main cause of exercise intolerance in individuals with hyperthyroidism is the change in energy metabolism. The number of studies investigating the exercise capacity in hyperthyroid patients is limited. Information support will be provided to the literature by evaluating the exercise capacity in patients with hyperthyroidism.

Physical activity is positively associated with changes in cardiovascular risk factors. Neuromuscular symptoms and exercise intolerance seen with thyroid hormone excess can lead people to an inactive life. Indirect calorimetry, the gold standard in energy expenditure, has been shown to be highly correlated with metabolic holter.There are no studies evaluating physical activity level with metabolic holter in individuals with hyperthyroidism. In this study, physical activity level will be evaluated by metabolic holter.

Patients with hyperthyroidism referred to the Cardiopulmonary Rehabilitation Unit of Gazi University Physiotherapy and Rehabilitation Department by the physicians of the Department of Endocrinology and Metabolism of the Department of Internal Diseases of Gazi University Faculty of Medicine will be included in the study. Patients and healthy individuals will be evaluated and the evaluation results will be compared. According to the sample size analysis 15 patients and 15 healthy individuals with similar demographic characteristics will be included the study. Patients and healthy individuals will be selected according to predetermined inclusion and exclusion criteria. Patients will be evaluated twice. The first evaluation will be made in the new diagnosis. The second evaluation will be made in the euthyroidism.The assessments will be completed in two days.

Functional exercise capacity (6 minutes walk test and 6 minutes stepper test), physical activity level (multi-sensor activity monitor), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), peripheral muscle strength (dynamometer), respiratory muscle endurance (incremental threshold loading test), quality of life (The Thyroid-Related Quality of Life-ThyPRO), fatigue (Fatigue Severity Scale), depression-anxiety-stress (Depression Anxiety Stress Scale-42), quality of sleep (Pittsburgh Sleep Quality Index) and shortness of breath (Modified Medical Research Council (MMRC)) will be evaluated.

ELIGIBILITY:
Inclusion criteria for patients group: Patients who are;

* Individuals diagnosed with hyperthyroidism by a physician
* Individuals between the ages of 18-70

Exclusion criteria for patients group: Patients who are;

* Use of drugs that affect the heart rate (except for short-term beta blockers given to relieve thyrotoxicosis symptoms)
* having problems that limit physical activity (orthopedic, neurological, psychological)
* having comorbidities such as uncontrolled hypertension, diabetes mellitus, heart failure or atrial fibrillation
* use of any medication that may affect thyroid function
* patients with acute infection during evaluation
* patients with uncontrolled hypertension, diabetes mellitus

Inclusion criteria for healthy group: Participants who are;

* being between ages of 18 and 70
* willing to participate to the study

Exclusion criteria for healthy group: Participants who are;

* having any diagnosis of chronic diseases
* having health problems such as cooperation
* having acute infection during evaluation
* being current smokers
* being ex-smokers (≥10 pack*years)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 15 patients with hyperthyroid will be included in patients group and 15 healthy individuals will be included in control group
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Functional Exercise Capacity | First Day
  Functional exercise capacity will be evaluated with 6-minutes walking test according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The total distance they walked for 6 minutes in a 30-meter straight corridor will be recorded.
Functional Exercise Capacity | Second Day
  Functional exercise capacity will be evaluated with 6-minutes Stepper Test according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The total number of steps will be recorded for 6 minutes.
Physical activity (Total energy expenditure) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Physical activity time (min / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Physical activity time (min / day)will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure (joule / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Active energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Average metabolic equivalent (MET / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Average metabolic equivalent (MET / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Number of steps (steps / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Number of steps (steps / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Time spent lying down (min / day) days)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Time spent lying down (min / day) days) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Sleep time (min / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Sleep time (min / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.

SECONDARY OUTCOMES:
Respiratory Muscle Strength | First Day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength will be measured with a portable mouth pressure measuring device according to ATS and ERS criteria.
Peripheral Muscle Strength | First Day
  Isometric peripheral muscle strength will be measured with a portable hand dynamometer (JTECH Commander, USA). Measurements will be repeated on the shoulder abductors and knee extensors three times on the right and left.
Respiratory Muscle Endurance | Second Day
  Respiratory muscle endurance will be assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd., Birmingham, UK) device and the respiratory muscle endurance test at increased threshold load. The test will be started with 20% of the maximal inspiratory pressure and the pressure will be increased to 40%, 60%, 80% and 100% every two minutes. Patients will be asked to continue breathing through the device during the test. During the test, the number of breaths delivered and the maximal time reached during each 2-minute period will be recorded. If the individual cannot breathe 3 consecutive times, the test will be terminated by the physiotherapist. The total duration of the test and the maximum pressure value at which it continues to breathe for at least 1 minute will be multiplied. The value found will be recorded as the respiratory muscle endurance value.inspiratory pressure with a 20% increment every 2 minutes.
Disease Specific Quality of Life | First Day
  Quality of life was evaluated with the Turkish version of the Quality of Life Scale (ThyPRO) in Thyroid Patients. For each question, a five-point Likert type (0 = not at all, 1 = very little, 2 = a little, 3 = a little bit, 4 = a lot) was used. Each subscale is scored differently. High scores indicate a decreased quality of life.
Fatigue | First Day
  Fatigue will be evaluated using Turkish version of Fatigue Severity Scale. This questionnaire includes 9 items and score range for each item from 1 to 7 point (7-point Likert scale). Fatigue Severity Scale score is calculates by deriving an arithmetic mean. Cut-scores of over 4 are indicative of significant fatigue (higher scores show more severe fatigue)score range for each item from 1 to 7 point (7-point Likert scale).
Shortness of breath | First Day
  The Modified Medical Research Council (MMRC) dyspnea scale will be used to determine the perception of dyspnea during activities of daily living.
  Dyspnea is graded as: zero (shortness of breath with strenuous exercise only); one (shortness of breath when rushing or walking up a slight uphill); two (because of shortness of breath they walk slower than people of the same age or have to stop to breathe while walking at their own pace); three (stops to breathe after walking 100 meters or after a few minutes); and four (too short of breath to leave the house or shortness of breath when getting dressed).daily living activities.
Sleep Quality | First Day
  Sleep quality will be evaluated by Turkish adaptation of Pittsburgh Sleep Quality Index (PSQI). The scale includes 24 questions. The questions included in the scoring consist of seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction. Total PSQI score varies between 0-21. A total score greater than five indicates "poor sleep quality".
Depression Anxiety Stress | First Day
  Depression, Anxiety and Stress Scale (DASS) was evaluated with Turkish version. The scale is a four-digit Likert type scale. The total scores of the scale vary between 0 and 42 for each sub-dimension. A high score indicates that the individual has that problem.
Pulmonary function (Forced vital capacity (FVC)) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society guidelines. Forced vital capacity (FVC) will be measured.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society guidelines. Forced expiratory volume in the first second (FEV1) will be measured.
Pulmonary function (FEV1 / FVC) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society guidelines. FEV1 / FVC will be measured.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society guidelines. Flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be measured.
Pulmonary function (Peak flow rate (PEF)) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society guidelines. Peak flow rate (PEF) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University; Fidan YILMAZ, Pt, Study Chair — Gazi University; Afruz BABAYEVA, MD, Principal Investigator — Gazi University; İlhan YETKİN, Prof. Dr., Principal Investigator — Gazi University
Locations (1):
- Gazi University Facutly of Health Sciences Department of Physiotheraphy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahaly G, Hellermann J, Mohr-Kahaly S, Treese N. Impaired cardiopulmonary exercise capacity in patients with hyperthyroidism. Chest. 1996 Jan;109(1):57-61. doi: 10.1378/chest.109.1.57. PMID 8549218
- [Background] Siafakas NM, Milona I, Salesiotou V, Filaditaki V, Tzanakis N, Bouros D. Respiratory muscle strength in hyperthyroidism before and after treatment. Am Rev Respir Dis. 1992 Oct;146(4):1025-9. doi: 10.1164/ajrccm/146.4.1025. PMID 1416391
- [Background] Goswami R, Guleria R, Gupta AK, Gupta N, Marwaha RK, Pande JN, Kochupillai N. Prevalence of diaphragmatic muscle weakness and dyspnoea in Graves' disease and their reversibility with carbimazole therapy. Eur J Endocrinol. 2002 Sep;147(3):299-303. doi: 10.1530/eje.0.1470299. PMID 12213666
- [Background] Kendrick AH, O'Reilly JF, Laszlo G. Lung function and exercise performance in hyperthyroidism before and after treatment. Q J Med. 1988 Aug;68(256):615-27. PMID 3255983
- [Background] McAllister RM, Delp MD, Laughlin MH. Thyroid status and exercise tolerance. Cardiovascular and metabolic considerations. Sports Med. 1995 Sep;20(3):189-98. doi: 10.2165/00007256-199520030-00005. PMID 8571001
- [Derived] Yilmaz F, Babayeva A, Yetkin I, Bosnak-Guclu M. Comparison of exercise capacity and physical activity in patients with hyperthyroidism and controls. J Bodyw Mov Ther. 2024 Oct;40:1752-1760. doi: 10.1016/j.jbmt.2024.10.029. Epub 2024 Oct 15. PMID 39593519